CLINICAL TRIAL: NCT04360434
Title: A Phase 1, First-in-Human, Double-Blind, Placebo-Controlled, Multicenter, Single and Multiple Ascending Dose Study of NI006 in Patients With Amyloid Transthyretin Cardiomyopathy Followed by an Open-Label Extension
Brief Title: First-in-Human Study of NI006 in Patients With Amyloid Transthyretin Cardiomyopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurimmune AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NI006-101; 2019-001932-80 (EudraCT Number)
Record Dates: First submitted 2020-03-11; First posted 2020-04-24 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Amyloid Transthyretin Cardiomyopathy
Keywords: ATTR; Transthyretin; Amyloidosis; Cardiomyopathy; ATTR-CM
MeSH Terms: conditions — Amyloidosis; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NI006 (Experimental): Dose escalation in up to 6 dose cohorts. Subjects will be administered a single dose of NI006 in the SAD, multiple doses of NI006 in the MAD and OLE phases.
  Interventions: Drug: NI006
- Placebo (Placebo Comparator): Subjects will be administered a single dose of placebo in the SAD phase and multiple doses of placebo in the MAD phase.
  In the OLE phase, all subjects will be administered multiple doses of NI006.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NI006 — NI006 will be administered intravenously
  Arms: NI006
Drug: Placebo — Formulation buffer of NI006, matching volume of NI006 doses will be administered intravenously
  Arms: Placebo

SUMMARY:
A phase 1, randomized, placebo-controlled, double-blind, dose escalation trial combining single-ascending dose and multiple-ascending dose phases of NI006 or placebo, followed by an open-label extension phase in subjects with Amyloid Transthyretin Cardiomyopathy (ATTR-CM).

DETAILED DESCRIPTION:
This phase 1, randomized, placebo-controlled, double-blind trial in subjects with Amyloid Transthyretin Cardiomyopathy (ATTR-CM) consists of single-ascending dose (SAD) and multiple-ascending dose (MAD) phases, followed by an open-label extension (OLE) phase.

In the SAD phase subjects are randomized in a 4:2 ratio to receive a single infusion of NI006 or placebo.

Subjects completing the SAD phase will be enrolled in the MAD phase upon evaluation of all available safety data and receive a maximum of 3 additional infusions of NI006 or placebo every 28 days.

Subjects completing the MAD phase will have the possibility to continue in an OLE phase with treatment up-titrations and switch from placebo to NI006 and receive up to 8 infusions of NI006 every 28 days.

Subjects of cohort 1 to 5 who received at least one dose of NI006 during the OLE phase will have the possibility for a second OLE phase (OLE2) after completing the OLE phase and receive up to 10 additional infusions of NI006 every 28 days.

In total, about 42 subjects are planned to be enrolled in 7 cohorts of 6 subjects each, at 6 ascending dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject prior to any trial-related procedure indicating that he/she understands the purpose of, and procedures required for the trial and is willing to participate in it
2. Male or female subjects aged ≥18 years (and < 85 years only for cohort 7) at the time of obtaining informed consent and with confirmed availability for the scheduled trial visits
3. Confirmed ATTR-Cardiomyopathy diagnosis established by:

   * Polarizing light microscopy of green birefringent material in Congo red-stained tissue specimens and confirmed diagnosis of ATTR amyloidosis by IHC or mass spectrometry OR
   * positive bone scintigraphy using either DPD, HMDP or PYP, with cardiac signal intensity indicative of ATTR-Cardiomyopathy (early phase imaging: cardiac mediastinum ratio > 1.21; late phase imaging: Perugini Grade 2 or 3) and absence of gammopathy (negative serum and urine immunofixation electrophoresis plus normal free light chain serum ratio). If a gammopathy is detected, diagnosis must be established based on tissue biopsy as indicated above
4. Known genotype as follows:

   1. Known pathogenic TTR mutation for subjects with hereditary ATTR- Cardiomyopathy
   2. Known negative genetic testing for a TTR mutation for subjects with sporadic, WT- ATTR-Cardiomyopathy
5. Chronic Heart Failure with all of the following characteristics:

   1. LVEF ≥40%
   2. LVWT ≥14 mm, measured by echocardiography
   3. NT-proBNP level ≥600 pg/mL
   4. Able to walk ≥150 meter in the 6-MWT
   5. NYHA class III (applicable only for cohort 7)
   6. No hospitalizations for cardiac disease for at least 30 calendar days prior to screening
6. General health status acceptable for a participation in a clinical trial with a Karnofsky Performance Status ≥60%
7. Stable pharmacological treatment of any other chronic condition for at least 30 calendar days prior to screening, with the exclusion of immunomodulatory and immunosuppressive treatments
8. ANC ≥1000 cells/mm³, platelet count ≥100,000 cells/mm³, and hemoglobin ≥10 g/dL
9. Women of childbearing potential must have a negative serum pregnancy test at screening and must agree to use highly effective physician-approved contraception from screening to 5 months after ending trial participation
10. Males must be surgically sterile or must agree to use highly effective physician-approved contraception throughout of the trial participation, and for 5 months after ending trial participation

Exclusion Criteria:

1. Amyloid light-chain amyloidosis or any other non ATTR amyloidosis
2. Heart failure corresponding to NYHA class IV
3. Uncontrolled hypertension with systolic pressure ≥180 mmHg or diastolic pressure ≥110 mmHg confirmed by 3 measurements in supine position recorded with 5 minutes break in between the measurements
4. Hypotension with systolic pressure ≤ 90 mmHg or diastolic pressure ≤ 60 mmHg confirmed by 3 measurements in supine position recorded with 5 minutes break in between the measurements
5. NT-proBNP ≥6'000 pg/mL (NT-proBNP ≥8'500 pg/mL applicable only for cohort 7)
6. Heart failure not predominantly caused by ATTR-Cardiomyopathy
7. Any severe uncorrected valve disease
8. Chronic liver disease with liver function test abnormalities:

   1. ALT and AST > 2.5 × ULN
   2. Total bilirubin > 2 × ULN
9. Respiratory insufficiency requiring oxygen therapy
10. Renal insufficiency with eGFR < 30 mL/min/1.73 m2 using the CKD-EPI equation
11. Active malignancy with exception of the following:

    1. Adequately treated basal cell carcinoma
    2. Squamous cell carcinoma of the skin
    3. In situ cervical cancer
    4. Low risk prostate cancer with Gleason score < 7 and prostate specific antigen < 10 mg/mL
    5. Any other cancer from which the subject has been disease-free for ≥ 2 years
12. Uncontrolled infection as per Investigator's judgement
13. Known HIV infection, seropositivity for HIV, hepatitis B and C as well as active hepatitis A
14. Autoimmune disease requiring immunosuppressive/modulating treatment in the last 2 years
15. History of organ transplantation or ventricular assist device
16. Polyneuropathy disability score > IIIA
17. Suspected or known intolerance/allergy to proteins or any components of the investigational medicinal product
18. Concomitant immunosuppressant therapy e.g., corticosteroids, prednisone, dexamethasone except as indicated in low dose (i.e., up to 10 mg prednisone or equivalent daily is allowed) for other medical conditions such as inhaled steroid for asthma
19. Use of the following drugs acting on TTR or ATTR: tolcapone, diflunisal, patisiran, inotersen, and long-term doxycycline, in the 30 calendar days prior to signing informed consent form. Tafamidis is permitted if it is given as standard of care in a stable dose for at least 30 calendar days prior to signing the informed consent form
20. Participation in another investigational clinical trial or intake of investigational drug within 30 calendar days before signing the informed consent form
21. Suspected or known drug or alcohol abuse
22. Serious psychiatric or any other medical condition (including laboratory abnormalities), which, in the opinion of the Investigator, makes the subject unsuitable for inclusion and puts the subject at an unacceptable risk
23. Subject is nursing or is considering becoming pregnant during the trial or in the 5 months after ending trial participation
24. Unwillingness or inability to adhere to the trial requirements
25. If subject is in any way dependent on Neurimmune AG or the principal Investigator or if the subject is accommodated in an establishment on judicial or administrative order
26. Employee or immediate family (spouse, parent, child or sibling, whether biological or legally adopted) of an employee of Neurimmune AG, the contract research organization or the trial site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Number and proportion of treatment emergent adverse events and serious adverse events and clinically significant changes in laboratory parameters, vital signs, electrocardiogram and echocardiogram | 4 months
  Number and proportion of treatment emergent adverse events and serious adverse events and clinically significant changes in laboratory parameters (hematology, clinical chemistry, immunology, urinalysis), vital signs, electrocardiogram and echocardiogram
Number and proportion of treatment emergent adverse events and serious adverse events and clinically significant changes in laboratory parameters, vital signs, electrocardiogram and echocardiogram | 12 months
  Number and proportion of treatment emergent adverse events and serious adverse events and clinically significant changes in laboratory parameters (hematology, clinical chemistry, immunology, urinalysis), vital signs, electrocardiogram and echocardiogram
Number and proportion of treatment emergent adverse events and serious adverse events and clinically significant changes in laboratory parameters, vital signs, electrocardiogram and echocardiogram | additional up to 10 months
  Number and proportion of treatment emergent adverse events and serious adverse events and clinically significant changes in laboratory parameters (hematology, clinical chemistry, immunology, urinalysis), vital signs, electrocardiogram and echocardiogram

SECONDARY OUTCOMES:
NI006 pharmacokinetic profile and parameters - Cmax | 4 months
  Maximum observed serum concentration (Cmax) of NI006
NI006 pharmacokinetic profile and parameters - Tmax | 4 months
  Time to maximum observed serum concentration (Tmax) of NI006
NI006 pharmacokinetic profile and parameters - AUCinf | 1 month
  Area under the serum concentration-time curve from zero to infinity (AUCinf) of NI006
NI006 pharmacokinetic profile and parameters - CL | 4 months
  Serum clearance (CL) of NI006
NI006 pharmacokinetic profile and parameters - Vz | 4 months
  NI006 apparent volume of distribution during terminal phase (Vz)
NI006 pharmacokinetic profile and parameters - Vss | 4 months
  NI006 apparent volume of distribution at steady state (Vss)
NI006 pharmacokinetic profile and parameters - t½ | 4 months
  Terminal elimination half-life (t½) of NI006 in serum
NI006 pharmacokinetic profile and parameters - AUCtau | 4 months
  Area under the serum concentration-time curve from time zero to the end of the dosing interval after the first dose (AUCtau) of NI006
NI006 pharmacokinetic profile and parameters - RaccCmax | 4 months
  Accumulation ratio for maximum concentration (RaccCmax) of NI006 in serum
NI006 pharmacokinetic profile and parameters - RaccAUC | 4 months
  Accumulation ratio calculated from AUC (RaccAUC) of NI006 in serum
NI006 pharmacokinetic profile and parameters - Ctrough | 12 months
  Minimum observed concentration (Ctrough) of NI006 in serum
NI006 OLE2 pharmacokinetic profile and parameters - Ctrough | up to 10 months
  Minimum observed concentration (Ctrough) of NI006 in serum
NI006 pharmacokinetic profile and parameters - dose-normalized Ctrough | 12 months
  Dose-normalized minimum observed concentration (Ctrough) of NI006 in serum
NI006 OLE2 pharmacokinetic profile and parameters - dose-normalized Ctrough | up to 10 months
  Dose-normalized minimum observed concentration (Ctrough) of NI006 in serum

OTHER OUTCOMES:
Exploratory - Efficacy of multiple doses of NI006 on 6-Minute Walk Test (6-MWT) | 4 and 12 months
  Changes in 6-MWT
Exploratory - Efficacy of multiple doses of NI006 on patient questionnaire outcome | 4 and 12 months
  Changes in patient questionnaire outcome
Exploratory - Efficacy of multiple doses of NI006 on amyloid load | 4 and 12 months
  Changes in amyloid load assessed by cardiac imaging
Exploratory - Efficacy of multiple doses of NI006 on cardiac biomarkers - NT-proBNP | 4 and 12 months
  Changes in NT-proBNP concentration
Exploratory - Efficacy of multiple doses of NI006 on cardiac biomarkers - Troponin-T | 4 and 12 months
  Changes in Troponin-T concentration
Exploratory - Immunogenicity of NI006 | 4 and 12 months
  Determination of anti-drug antibody response

CONTACTS AND LOCATIONS:
Locations (6):
- France (3):
  - Hôpital Henri Mondor, Créteil
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU Toulouse - Hôpital Rangueil, Toulouse
- Universitätsklinikum Heidelberg, Heidelberg, Germany
- University Medical Center Groningen, Groningen, Netherlands
- Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia-Pavia P, Aus dem Siepen F, Donal E, Lairez O, van der Meer P, Kristen AV, Mercuri MF, Michalon A, Frost RJA, Grimm J, Nitsch RM, Hock C, Kahr PC, Damy T. Phase 1 Trial of Antibody NI006 for Depletion of Cardiac Transthyretin Amyloid. N Engl J Med. 2023 Jul 20;389(3):239-250. doi: 10.1056/NEJMoa2303765. Epub 2023 May 20. PMID 37212440